CLINICAL TRIAL: NCT07242001
Title: The Effectiveness of Laser Acupuncture in the Management of Otitis Media With Effusion in Children
Brief Title: Laser Acupuncture for Otitis Media With Effusion in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Agitha Melita Putri, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-09-1474
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Otitis Media With Effusion
MeSH Terms: conditions — Otitis Media with Effusion

STUDY DESIGN:
Intervention Model Description: The treatment group receiving active laser acupuncture and standard decongestants while the control group receiving sham laser acupuncture and standard decongestants.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding will be applied to participants and outcome assessors. Group allocation will not be disclosed to them to minimize assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Active laser acupuncture and standard decongestants.
  Interventions: Device: Laser Acupuncture
- Control Group (Sham Comparator): Sham laser acupuncture and standard decongestants.
  Interventions: Device: Sham Laser Acupuncture

INTERVENTIONS:
Device: Laser Acupuncture — Laser Acupuncture is performed for 40 seconds per point at acupoints SI19, TE17, TE5, and LI4 using a low-level laser device (785 nm, 50 mW, delivering an energy density of 12.73 J/cm²). The device is activated to emit laser energy. Standard aseptic procedures are followed. The laser applicator is held perpendicular to the skin without pressure. Participants continue their routine decongestant therapy.
  Arms: Intervention Group
Device: Sham Laser Acupuncture — Sham Laser Acupuncture involves placing the applicator of an inactive laser device onto the same acupoints (SI19, TE17, TE5, and LI4) for the same duration as the active group. The device is turned on, but the start button is not pressed, so no laser energy is emitted. All procedures, including aseptic preparation, timing, and handling of the device, are performed identically to the intervention group to maintain blinding. Participants will wear ear covers and the device's LCD panel will be covered. Participants continue their routine decongestant therapy.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to learn if laser acupuncture (LA) can improve middle ear function and reduce the recurrence of Otitis Media with Effusion (OME) in children. The main questions it aims to answer are:

Does LA, when combined with standard treatment (decongestants), improve middle ear function as measured by tympanometry immediately after the 2-week intervention? Does LA, when combined with standard treatment, reduce the recurrence rate of OME as monitored over a 1-month period after the intervention? What is the safety profile of LA in this population, as measured by the incidence of adverse events? Researchers will compare active LA to sham LA (a placebo procedure with an inactive device) to determine if LA leads to meaningful improvements in children with OME.

Participants will:

Complete an initial assessment using tympanometry to confirm the diagnosis. Receive four sessions of either active LA or sham LA over a 2-week period. Complete a final assessment using tympanometry after the final session. Participate in a 1-month follow-up period with weekly monitoring for recurrence.

DETAILED DESCRIPTION:
This is a double-blind, randomized controlled trial designed to assess the effectiveness and safety of laser acupuncture as an adjunctive therapy for Otitis Media with Effusion (OME) in children. A total of 32 participants aged 2-10 years will be randomly assigned to either a treatment group (receiving active laser acupuncture and standard decongestants) or a control group (receiving sham laser acupuncture and standard decongestants). The intervention consists of four sessions over two weeks. The primary outcome is the improvement of middle ear function, measured by a change in tympanometry results from Type B to Type A. Secondary outcomes include the rate of OME recurrence at one month and the incidence of adverse events during the therapy period. This study will provide evidence on whether laser acupuncture is a beneficial, non-invasive treatment option for this common pediatric condition.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-10 years, both male and female.
* Diagnosed with OME with a Type B tympanogram curve, either unilateral or bilateral.
* No acute ear infection within the last 2 weeks.
* Willingness to participate in the study until completion and signed informed consent from a parent or legal guardian.

Exclusion Criteria:

* History of tympanic membrane perforation or previous ear surgery.
* Presence of severe OME complications, such as permanent hearing loss, tympanosclerosis, or cholesteatoma.
* Underwent laser acupuncture therapy for OME within the last three months.
* History of unstable systemic disease or other medical conditions that could interfere with the study, such as a history of uncontrolled seizures or epilepsy, a current high fever >38°C, or malignancy/cancer in the ENT system.
* Presence of a mental disorder, inability to communicate well, or being uncooperative.
* Presence of wounds or skin lesions at the intended acupuncture point irradiation sites.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Tympanogram Results | Baseline and immediately after the final (4th) therapy session at 2 weeks.
  Improvement in middle ear function will be assessed using tympanometry. The outcome is measured as the proportion of participants whose tympanogram curve change from Type B (indicating effusion) to Type A (normal).

SECONDARY OUTCOMES:
Recurrence Rate of OME | From the end of the intervention over a 1-month follow-up period.
  The number of participants who experience a recurrence of OME symptoms after the intervention period will be recorded, assessed via weekly monitoring.
Time to First Recurrence | From the end of the intervention over a 1-month follow-up period.
  ime (in days/weeks) from the end of the intervention to the first documented recurrence of OME will be measured.
Incidence of Adverse Events | At the end of each of the four acupuncture therapy sessions.
  The total number, type, and severity of adverse events reported by participants will be documented throughout the therapy period.

CONTACTS AND LOCATIONS:
Overall Officials: KPEK FKUI-RSCM, Principal Investigator — The Health Research Ethics Commitee - Faculty of Medicine Universitas Indonesia and Dr. Cipto Mangunkusumo National Hospital
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No